CLINICAL TRIAL: NCT04985630
Title: Open-labelled Study to Validate Home-based Use of a Health and Wellness Kit (The Mitopure Challenge) to Detect Levels of Urolithin A in Dried Blood Spots After Intake of Mitopure (Proprietary Urolithin A)
Brief Title: The Mitopure Challenge to Detect Levels of Urolithin A in Dried Blood Spots
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amazentis SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 21.02.AMZ
Record Dates: First submitted 2021-07-13; First posted 2021-08-02 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Healthy Aging; Healthy; Healthy Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mitopure Challenge to assess blood levels of Urolithin A after dietary and Mitopure intake (Experimental): Mitopure challenge with diet (Pomegranate juice- Before) followed by Mitopure supplementation (After) to compare levels in blood spots of UA-Glucuronide (in ng/mL)
  Interventions: Dietary Supplement: Mitopure; Dietary Supplement: Pomegranate Juice

INTERVENTIONS:
Dietary Supplement: Mitopure — Fruit flavored sachet containing fixed dose of Mitopure™ (Proprietary Urolithin A)
Dietary Supplement: Pomegranate Juice — 100% Pomegranate juice

SUMMARY:
Open labelled, virtual home based study to assess the test repeatability and the failure/rejection rate of the samples collected at home by participants.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18 to 80 years of age;
2. Is in general good health, as determined by the research team;
3. Willingness to consume the investigation product, complete questionnaires and to complete the study;
4. Have given voluntary, electronic, informed consent to be a participant in the study.

Exclusion Criteria:

1. Women who are pregnant, breastfeeding, or planning to become pregnant during the course of the trial;
2. Volunteers who plan to donate blood during the study or within 30 days of completing the study;
3. Subject has a known allergy to the test material's active or inactive ingredients;
4. Subjects with unstable medical conditions;
5. Participation in a clinical research trial within 30 days prior to randomization;
6. Allergy or sensitivity to study ingredients;
7. Individuals who are cognitively impaired and/or who are unable to give informed consent;
8. Any other condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject;
9. Has taken antibiotics within the previous 30 days.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2021-08-30 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Failure/rejection rate (% of the samples) collected at home by participants. | 4 weeks
  Acceptability target goal is to hit 80% of analyzed samples

SECONDARY OUTCOMES:
Sensitivity and specificity (% of the samples) of the analytical method developed to test Urolithin A in dry blood spots. | 4 weeks
Fold change increase in the levels of UA-Glucuronide (in ng/mL) in the dried blood spots provided in the kit before and after the challenge | 4 weeks
Validation of a health questionnaire on participants health status | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anurag Singh, MD, PhD, Principal Investigator — Amazentis SA
Locations (1):
- Amazentis USA, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singh A, D'Amico D, Andreux PA, Dunngalvin G, Kern T, Blanco-Bose W, Auwerx J, Aebischer P, Rinsch C. Direct supplementation with Urolithin A overcomes limitations of dietary exposure and gut microbiome variability in healthy adults to achieve consistent levels across the population. Eur J Clin Nutr. 2022 Feb;76(2):297-308. doi: 10.1038/s41430-021-00950-1. Epub 2021 Jun 11. PMID 34117375